CLINICAL TRIAL: NCT01677637
Title: Epidemiological, Observational, Multicenter Clinical Trial
Brief Title: Osteoporosis Screening Trial
Acronym: OSTRIA
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-BOD-EL-02
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2013-05

CONDITIONS: Osteoporosis
Keywords: osteopenia, postmenopausal
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All measurements: Total measured population

SUMMARY:
Osteoporosis is the most common disease of bone and characterized firstly by low bone mass and secondly, impaired bone microarchitecture structure resulting in reduced strength and increased risk of fracture. Osteoporosis is divided into: primary (Postmenopausal Osteoporosis Osteoporosis & elderly and senile osteoporosis) and secondary. The most common form is postmenopausal osteoporosis. It occurs in women after menopause and is associated with decreased estrogen production, which normally occurs at this age women Osteoporosis usually occurs after age 50, it is very common in women than in men, and its frequency increases with advancing age.

DETAILED DESCRIPTION:
According to the findings of epidemiological studies in different countries, osteoporosis affects 25-35% of women and 15-20% of men aged 50 and over. In terms of our country in the recent nation-epidemiological research on rheumatic diseases in the general adult population, ie persons aged 19 and over, organized and conducted by the Greek Institute of Rheumatology Research, became a separate study on frequency of osteoporosis in women aged 50 years and above. These women was measured BMD at the lumbar spine and at the upper end of the femur and found that 28.4% of Greek women aged 50 and over have osteoporosis. It is indeed very interesting finding in this study that women who have osteoporosis, the vast majority, ie about 75%, I do not know. This is of particular importance and highlights the need to educate and inform systematically the public, especially women regarding both the modern possibilities for early diagnosis of osteoporosis, and for the implementation of primary and secondary prevention.

Osteoporosis is a major public health problem for two reasons: First, because it is common, and secondly because it has significant impact on patients and their families, the health system and the national economy.

The main clinical manifestation of osteoporosis is fractures low energy, ie fractures occurring after mild degree injury, eg fall from a standing position. Approximately 40% of cases osteoporotic fractures on the vertebrae, 20% in the femoral neck, 20% to 20% radius and several other bones. While osteoporosis is generally regarded as a disease of women, however, as already mentioned above, osteoporosis affects and men. It has even been found that 30% of osteoporotic fractures of the femoral neck and 20% of osteoporotic vertebral fractures occur in men.

The risk of fractures of the hip, vertebrae and radius increases with advancing age in both women and men. It has even been estimated that the risk of osteoporotic fracture in women aged 50 and over is 40-50% and 15-20% in men.

The adverse effects of osteoporosis patients and their families, the health system and the national economy due to fractures. Indicative only some of these effects:

* The mortality in patients with hip fractures and clinically symptomatic vertebral fractures is significantly higher than that observed in individuals of the same sex and similar age in the general population. For example, within the first year after the fracture approximately 20% of patients with hip fracture and 25% of patients with vertebral fracture die.
* One year after a hip fracture, only 50% of patients can execute without help ordinary activities of everyday life.
* On an annual basis the number of days of hospitalization for patients with osteoporotic fractures is significantly greater than the number of days of hospitalization required for patients with stroke or diabetes mellitus or myocardial infarction or breast cancer.

Moreover, in 2000 the European Union the then 15 Member States (total population of 379,000,000 people) is estimated to have occurred 3.79 million osteoporotic fractures and that the direct costs of these fractures (costs of hospitalization, surgery and medical care) was approximately 32 billion Euros.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Postmenopausal women
* Outpatients screened for osteoporosis
* Women > 45 years
* Women < 45 years under menopause
* Women obtained their consent to be measured

Exclusion Criteria:

* Premenopausal females
* Women without any symptom of menopause
* Women not obtained their consent to be measured

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal females screened for osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Osteoporosis Indicator | 1 year
  T-score per female as measured by Holofic Sahara Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Aristeidis Kerasiotis, Endocrinologist, Study Chair — Director of Endocrinology Unit ,'Iaso' Hospital of Athens, 37-39 Kifisias avenue, 15123, Athens, Greece; Ioannis Lentzas, MD, Principal Investigator — Director, Medical State Center, Simopoulo, Perfecture of Ilia; Dimitrios Tsorntanidis, MD, Principal Investigator — Registrat B', Medical State Center, Erymantheia, Achaia Perfecture; Maria Chronopoulou, MD, Principal Investigator — Registrat B', Medical State Site, Diakofto, Achaia Perfecture; Olimpia Raftopoulou, MD, Principal Investigator — Registrat B', Medical State Site, Myrsini, Perfecture of Ilia; Stylianos Danelakis, GP, Principal Investigator — Medical State Site, Leontari; Thomas Simos, GP, Principal Investigator — Medical State Site, Anavra; Theofanis Tsirogiannis, GP, Principal Investigator — Medical State Site, Agnantero; Konstantinos Vatalis, GP, Principal Investigator — Medical State Site, Tsartsani; Ioannis Antonopoulos, GP, Principal Investigator — Medical State Site, Ampelonas; Labros Kontovos, GP, Principal Investigator — Medical State Site, Nikaia, Perfecture of Larisa; Chara Kalliora, GP, Principal Investigator — Medical State Site, Gomfon, Perfecture of Trikala; Athanasios Misios, GP, Principal Investigator — Medical State Site, Megala Kalyvia; Antonis Monastiriotis, GP, Principal Investigator — Medical State Site, Oropos - Chalkoutsi; Zeppos Monstratos, GP, Principal Investigator — Medical State Site, Marathonas; George Sakellaropoulos, Orthop., Principal Investigator — Medical State Site, Marathonas; Andreas Sotiriou, Orthop., Principal Investigator — Private Office, Zografou, Athens; Maria Degaiti, GP, Principal Investigator — Medical State Site, Ano Mera, Island of Mykonos; Aristeidis Frydas, Medical Internist, Principal Investigator — Director, Medical State Center, Plomari, Island of Lesvos; Nikolaos Tsamouras, GP, Principal Investigator — Medical State Center, Agiassos, Island of Lesvos; Ioannis Komninos, GP, Principal Investigator — Medical State Center of Neapolis; Nikolaos Tsakountakis, GP, Principal Investigator — Medical State Center of Kastelli, Creta Island; Emmanouel Paterakis, GP, Principal Investigator — Private Madical Office, Heraklion, Creta Island; Panagiota Gourgoulia, MD, Principal Investigator — Regional State Medical Center of Giannouli - Tyrnavos, Perfecture of Larisa, Greece; Zisis Kelepouris, GP, Principal Investigator — Regional State Medical Center Platanos-Raxa, Perfecture of Trikala, Greece; Christos Ganochoritis, GP, Principal Investigator — Medical State Center of Pyrgetos and Egani, Regional Perfecture of Larisa; Demetra Zambouka, GP, Principal Investigator — Medical State Center of Agioi Anargyri, Regional Perfecture of Larisa; Charalampos Terzopoulos, MD, Orthopedics, Principal Investigator — Private office, Zografou, Athens, Greece; John Sakellariou, MD, Pathology, Registrat A, Principal Investigator — Medical Center of Farkadona, Thessalia, Greece; Aglaia Roganaki, MD, Registrat B,, Principal Investigator — Peripheral Medical Center of Mitropolis, Thessalia, Greece; Vasilis Delezos, MD, Registrat B, Principal Investigator — Medical Center of Sophades, Thessalia, Greece; Victoria Katsouri, MD, Registrat B, Principal Investigator — Medical Center of Sophades, Thessalia, Greece; Maria Papala, MD, Principal Investigator — State Medical Center of Tyrnavos, Thessalia, Greece; Styliani Papakosta, MD, Phyciatry, Principal Investigator — Medical Private Office, Larisa, Greece; Athanasios Tsivgoulis, MD in Physiatry, Principal Investigator — Medical Diagnosis Center, Lesvos Island, Greece; Petros Prokopis, MD, Principal Investigator — Medical Office of Avlona; George Papadimitriou, MD, Orthopedics, Principal Investigator — Private Medical Office, Vari Attikis; Vasilios Hamos, MD, Director, Principal Investigator — State Medical Cener, Agia, Larissa; Lemonia Arvanitakou, MD, Principal Investigator — State Medical Center, Agia, Larissa; Victoria Rizou, MD, Principal Investigator — State Medical Office, Halki, Larissa; Vassiliki Mamakou, MD, Internist, Principal Investigator — Mytilini; Antonios Partsinevelos, MD, Orth, Principal Investigator — Private Office, Marousi, Athens; George Patoulis, MD, Orth, Principal Investigator — Private Office, Marousi, Athens
Locations (1):
- Iaso Hospital of Athens, Center of Endocrinology and Bone Metabolism, Athens, Kifisias Avenue, 37-39, Maroussi, Greece

REFERENCES:
- [Background] Kanis JA. Assessment of fracture risk and its application to screening for postmenopausal osteoporosis: synopsis of a WHO report. WHO Study Group. Osteoporos Int. 1994 Nov;4(6):368-81. doi: 10.1007/BF01622200. PMID 7696835
- [Background] McClung M. Difference in Distribution of T-scores Among Bone Density Tests in Postmenopausal Women. Bone Vol. 23, (5S), pg. S193, 1998.
- [Background] Ikeda Y, Iki M, Morita A, Aihara H, Kagamimori S, Kagawa Y, Matsuzaki T, Yoneshima H, Marumo F; JPOS Study Group. Age-specific values and cutoff levels for the diagnosis of osteoporosis in quantitative ultrasound measurements at the calcaneus with SAHARA in healthy Japanese women: Japanese population-based osteoporosis (JPOS) study. Calcif Tissue Int. 2002 Jul;71(1):1-9. doi: 10.1007/s00223-001-2079-6. Epub 2002 Jun 20. PMID 12200654
- [Background] Magkos F, Manios Y, Babaroutsi E, Sidossis LS. Quantitative ultrasound calcaneus measurements: normative data for the Greek population. Osteoporos Int. 2005 Mar;16(3):280-8. doi: 10.1007/s00198-004-1670-x. Epub 2004 Jul 6. PMID 15241583